CLINICAL TRIAL: NCT05219747
Title: The Effectiveness and Safety of Mucoadhesive Film Containing Acmella Oleracea Extract in Healthy Subjects: A Randomized Control Trial
Brief Title: The Effectiveness and Safety of Mucoadhesive Film Containing A.Oleracea Extract
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Kemporn Kitsahawong, Associated professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KKUHE641398
Record Dates: First submitted 2021-12-01; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2021-12

CONDITIONS: Oral Mucosa
Keywords: Mucoadhesive

STUDY DESIGN:
Intervention Model Description: Randomize control trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A.Oleracea group (Experimental): Mucoadhesive film containing Acmella oleracea extract
  Interventions: Other: Mucoadhesive film containing Acmella oleracea extract
- Placebo group (Placebo Comparator): Mucoadhesive film without Acmella oleracea extract
  Interventions: Other: Mucoadhesive film without Acmella oleracea extract

INTERVENTIONS:
Other: Mucoadhesive film containing Acmella oleracea extract — Participants will apply a mucoadhesive film containing Acmella oleracea extract on labial mucosa of lower lip by themselves at least for 2 hours
  Arms: A.Oleracea group
Other: Mucoadhesive film without Acmella oleracea extract — Participants will apply a mucoadhesive film on labial mucosa of lower lip by themselves at least for 2 hours
  Arms: Placebo group

SUMMARY:
Several natural products have been use to promote wound healing and relieve pain. Acmella oleracea has a component that has anesthetic and anti-inflammatory properties.

The mucoadhesive film can be improved by drug delivery system due to close contact with the absorption tissue leading to improvement in both local and systemic effects.

This study aims to evaluate the effectiveness and safety of mucoadhesive film containing Acmella oleracea extract in healthy subjects. This is a randomised, double-blind (participant and investigator), parallel-controlled clinical trial. In total, approximately 72 subjects will be enrolled into study.

Objectives

1. To investigate the potential of skin allergy reaction to mucoadhesive film containing Acmella oleracea extract in healthy subjects
2. To study the duration of mucosal adhesion of mucoadhesive film
3. To study the local anesthetic effect, participant's satisfaction and adverse effect of mucoadhesive film containing Acmella oleracea extract

DETAILED DESCRIPTION:
Total 72 Participants will divided into 2 groups by dentist who was not an examiner performed the randomization using blocked randomization (block of 4) from program of https://www.sealedenvelope.com/simple-randomiser/v1/lists/1. Study group will receive mucoadhesive film containing Acmella oleracea extract while control group will receive mucoadhesive film without active component. All participants in the study group will be test for allergic reaction of mucoadhesive film by skin prick test and patch skin test before testing and have to follow-up appointments (at 2, 4 and 7 days after skin test). At first visit, all participants will received oral examination and informed how to use mucoadhesive film by examiner. Then participants will asked to apply the mucoadhesive film at oral mucosa of lower lip. The effectiveness of intra-oral mucoadhesive film in this study will evaluated as follows :

1. Duration of mucosal adhesion and adverse effect by self report
2. The local anesthetic effect by using Numeric rating scale (NRS)
3. Participant's satisfaction by using Numeric rating scale (NRS)

The statistical methods :

General and oral health data, duration of mucosal adhesion will reported as frequencies, percentages and means (Standard deviation). The different of NRS score between groups will analyzed Independent t- test or Mann-Whitney U test. Using SPSS software. Statistically significant will considered at p-value < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy people age 18-60 years old and do not have regular medication.
2. Able to give the consent formation in a study and to cooperate in answering questionnaires or data records in google formation.
3. The participants must not have any wounds, tattoos, inflammation or pathology on the oral mucosa and skin of testing area.
4. The participants who can come to follow up for a specified period of time.

Exclusion Criteria:

1. The participants who need dental treatment or necessary to use topical medication to treat oral diseases during the study period (7 days).
2. History of allergic to the components of mucoadhesive film and/or have a history of other allergies.
3. The vulnerable participants include pregnancy or lactating women and disabilities.
4. History of using antihistamines drugs during the one-week period prior to joining the study or participants who need to use such antihistamines during the time participating in the study.
5. History of using topical gluco-corticosteroids during the one-week period on skin testing areas.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-02-28 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
To investigate the potential of skin allergy reaction to mucoadhesive film containing Acmella oleracea extract by skin prick test | Evaluate at 15 minutes after test in the 1st visit
  Outcome will be a number of participants with skin allergic reaction assessed by skin prick test
To investigate the potential of skin allergy reaction to mucoadhesive film containing Acmella oleracea extract by patch skin test at 2nd day after test | Evaluate at 2 days after patch skin test application
  Outcome will be a number of participants with skin allergic reaction assessed by patch skin test at 2nd day after test
To investigate the potential of skin allergy reaction to mucoadhesive film containing Acmella oleracea extract by patch skin test at 4th day after test | Evaluate at 4th day after patch skin test application
  Outcome will be a number of participants with skin allergic reaction assessed by path skin test at 4th day after test.
To investigate the potential of skin allergy reaction to mucoadhesive film containing Acmella oleracea extract by patch skin test at 7th day after test | Evaluate at 7th day after patch skin test application
  Outcome will be a number of participants with skin allergic reaction assessed by path skin test at 7th day after test.
To study the duration of mucosal adhesion of mucoadhesive film in healthy oral mucosa | Self reporting the time at which the film detaches (e.g. 16.30 hr.), within 24 hours after mucoadhesive film application
  Outcomes will be the duration in minutes of the mucoadhesive film adhering to participant' s oral mucosa
To study the local anesthetic effect | Self reporting at 1st visit, at 3 and 5minutes after application
  Outcome will be a score of Numeric rating scale (NRS) of local anesthetic effect. On a scale of 0-10, where 0 = no anesthetic effect and 10 = completely anesthetize
To study adverse effect related to mucoadhesive film use | Evaluate within 2 hours after mucoadhesive film application
  Outcome will be a number of participants who have adverse effect and the symptom of adverse effect
To evaluate participant's satisfaction | Evaluate at 2 hours after mucoadhesive film application
  Outcome will be a score of Numeric rating scale (NRS) of satisfaction of mucoadhesive film use. On a scale of 0-10, where 0 = totally unsatisfied and 10 = the most satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Kemporn Kitsahawong, DDS,MSc,PhD, Principal Investigator — Faculty of Dentistry, Khon Kaen University
Locations (1):
- Faculty of Dentistry , Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No